CLINICAL TRIAL: NCT01932749
Title: The Comparison of Effectiveness of Bilateral rTMS Versus Unilateral TMS in Patients With Bipolar Depression: a Study Randomized and Single Blind
Brief Title: The Study of Effectiveness Repetitive Transcranial Magnetic Stimulation in Bipolar Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tehran (Other)
Responsible Party: Principal Investigator, reza kazemi, Researcher, The Neuroscience Center, LLC
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 143
Record Dates: First submitted 2013-08-22; First posted 2013-08-30 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bilateral repetitive transcranial magnetic stimulation (Active Comparator): Bilateral protocol:
  Motor threshold 100% /LDLPFC/10Hz/5 second duration/10 second intertrain/ Motor threshold 120% /RDLPFC/1Hz/10 second duration/2second intertrain/
  Interventions: Device: Transcranial Magnetic stimulation
- unilateral repetitive transcranial magnetic stimulation (Active Comparator): Unilateral protocol:
  Motor threshold 120% /RDLPFC/1Hz/10 second duration/2second intertrain
  Interventions: Device: Transcranial Magnetic stimulation

INTERVENTIONS:
Device: Transcranial Magnetic stimulation
  Other Names: Magstim rapid 2

SUMMARY:
The aim of this study is to investigate the effect of repetitive TMS in reduction of depressive symptoms in patients with bipolar disorder. In a randomized, single blind clinical trials, 30 patients with bipolar disorder in Atieh Neuroscience center will be assigned to receive bilateral TMS and unilateral TMS, daily; for 20 sessions. The depressive and anxiety symptoms and quality of life will be assessed before the treatment (pre test) during the treatment (10th session), and after the treatment (post test). QEEG apply before and after rTMS in all subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients male and female with the range of 18-65 years of age
2. The diagnosis of Bipolar disorder according to DSM-IV-TR
3. Completion of consent form
4. Being under supervision of a psychiatrist,
5. Having BDI>14
6. Being able to adhere to treatment schedule,
7. Having stable symptoms as defined by not requiring a change in medication for at least 4 weeks .

Exclusion Criteria:

1. The history of rTMS treatment for any reason
2. Intracranial implant and other ferromagnetic materials close to the head
3. Cardiac pacemaker
4. Drug pumps
5. The risk of seizure with any reasons
6. High intracranial pressure
7. The history of epilepsy or seizure in the first relatives
8. Any metal in head
9. Pregnancy
10. Breastfeeding
11. High risk of suicide 12 Having personality disorder in axis II

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-08; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in depression severity.Depression will be assessed using the Beck depression inventory | Baseline to four weeks
  The BDI-II is measured depressive symptoms is administered before treatment, session 10, immediately after treatment.

SECONDARY OUTCOMES:
Change in anxiety severity .Anxiety will be assessed using the Beck Anxiety inventory. | Test Day 1, 10 & 20
  The BAI is measured for anxiety and is administered before treatment, session 10, immediately after treatment.
Change in World Health Organization Quality of Life- BREF (WHOQOL-BREF) | Test Day 1, 10& 20
  The WHOQOL-BREF is administered for measuring of quality of life before treatment, session 10, immediately after treatment
Change in QEEG and low resolution brain electromagnetic tomography (LORETA) | Before treatment, immediately after treatment
  QEEG and LORETA is applying for assessment brain waves patterns

CONTACTS AND LOCATIONS:
Locations (1):
- Atieh neuroscience center, Tehran, Tehran Province, Iran